CLINICAL TRIAL: NCT02099578
Title: Daily Incorporation of Strawberries Into a Diet Favorably Improves Vascular Function and Lowers Aortic Blood Pressure in Postmenopausal Women With Prehypertension
Brief Title: The Effects of Strawberries on Blood Pressure in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Principal Investigator, Bahram Arjmandi, Margaret A. Sitton Professor and Director of the Center for Advancing Exercise and Nutrition Research on Aging, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2013.11762
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
Keywords: Blood pressure; Arterial stiffness; Pulse wave velocity; Strawberries; Endothelial function; Oxidative stress; Postmenopausal women
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Freeze-dried placebo powder - two doses of 25 g/day for 8 weeks
  Interventions: Dietary Supplement: Placebo Powder
- 25 g of Freeze-dried Strawberry Powder (Active Comparator): Freeze-dried strawberry and placebo powder - one dose of 25 g/day of each for 8 weeks
  Interventions: Dietary Supplement: 25 g of Freeze-dried Strawberry Powder; Dietary Supplement: Placebo Powder
- 50 g of Freeze-dried Strawberry Powder (Experimental): Freeze-dried strawberry powder - two doses of 25 g/day for 8 weeks
  Interventions: Dietary Supplement: 50 g of Freeze-dried Strawberry Powder

INTERVENTIONS:
Dietary Supplement: 25 g of Freeze-dried Strawberry Powder — Participants will be given one packet of 25 g of freeze-dried strawberry powder and one packet of 25 g of placebo powder and asked to consume one packet in the morning and one at night.
  Other Names: California Strawberry Commission
  Arms: 25 g of Freeze-dried Strawberry Powder
Dietary Supplement: 50 g of Freeze-dried Strawberry Powder — Participants will be given two packets of 25 g of freeze-dried strawberry powder and asked to consume one packet in the morning and one at night.
  Other Names: California Strawberry Commission
  Arms: 50 g of Freeze-dried Strawberry Powder
Dietary Supplement: Placebo Powder — Participants will be given two packets of 25 g of placebo powder and asked to consume one packet in the morning and one at night.
  Other Names: California Strawberry Commission
  Arms: 25 g of Freeze-dried Strawberry Powder; Control Group

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the US. Statistics show that approximately 91% of individuals with CVD have vascular dysfunction. Hypertension is a major modifiable risk factor for CVD and approximately 60% of adults in the US are pre-hypertensive and hypertensive. In addition, the prevalence of hypertension is associated with aging in both genders; however, the increase in blood pressure (BP) in women after menopause exceeds that of men.

The development of effective and safe strategies to improve vascular function is of significance as it can have a great impact on quality of life, productivity and economic burden for the affected populations. One such alternative would be to introduce into the diet food sources that are rich in naturally occurring bioactive compounds. Thus, the long-term goal of the investigators is to provide feasible and effective dietary ways for postmenopausal women to improve their vascular function and quality of life.

Strawberries are a rich source of bioactive compounds and its total antioxidant content ranks third among all fruits and vegetables. Hence, the purpose of this study is to bring forth evidence that incorporation of strawberries into the diet will reduce blood pressure and improve cardiovascular function in pre- and stage 1-hypertensive postmenopausal women.

Sixty eligible postmenopausal women between the ages of 45 and 65 and a seated BP of ≥ 130/85 mm Hg but ≤ 160/100 mmHg at the screening visit will be randomly assigned to one of three groups:

1. 25 g freeze-dried strawberry powder;
2. 50 g freeze-dried strawberry powder; or
3. placebo powder. Participants will be asked to consume the supplements for 8-weeks. Medical history, medication use, dietary intake, and physical activity will be assessed at 0-, 4-, and 8-weeks followed by blood draw. Serum levels of markers of cardiovascular function as well as oxidative stress and inflammation will be measured.

The investigators hypothesize that regular consumption of strawberry will improve cardiovascular function, decrease BP and blood markers of oxidative stress as well as inflammation. Investigators also expect the findings of this study to provide a foundation for further studies to examine the effects of long-term incorporation of strawberry into the diet and the integrity of cardiovascular system.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (1 to 10 years after natural menopause or bilateral oophorectomy)
* 45-65 years of age
* Seated blood pressure ≥ 130/85 mm Hg but ≤ 160/100 mm Hg
* BMI > 25 but < 40 kg/m2

Exclusion Criteria:

* Seated blood pressure ≤ 129/84 or ≥160/101 mmHg
* Type I Diabetes
* Cardiovascular disease
* Active cancer
* Glaucoma
* Thyroid disease
* Kidney disease
* Liver disease
* Pancreatic disease
* Enrollment in a weight loss program
* Heavy smokers (>20 cigarettes per day)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8 weeks
  By measuring blood pressure variability and baroreflex sensitivity at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).

SECONDARY OUTCOMES:
Arterial Stiffness | 8 weeks
  By assessing pulse wave velocity and augmentation index at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).
Endothelial function | 8 weeks
  By assessing blood biomarkers of vascular function (adiponectin, leptin, endothelin-1, angiotensin II and 8-isoprostane).
Oxidative Stress | 8 weeks
  By assessing blood biomarkers of oxidative stress (superoxide dismutase, nitrate/nitrite, 8-isoprostane, malondialdehyde , and oxidized low density lipoprotein).
Inflammation | 8 weeks
  By assessing blood biomarkers of inflammation (tumor necrosis factor-α and C-reactive protein).

CONTACTS AND LOCATIONS:
Overall Officials: Bahram H Arjmandi, PhD, RD, Principal Investigator — Florida State University; Arturo Figueroa, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feresin RG, Johnson SA, Pourafshar S, Campbell JC, Jaime SJ, Navaei N, Elam ML, Akhavan NS, Alvarez-Alvarado S, Tenenbaum G, Brummel-Smith K, Salazar G, Figueroa A, Arjmandi BH. Impact of daily strawberry consumption on blood pressure and arterial stiffness in pre- and stage 1-hypertensive postmenopausal women: a randomized controlled trial. Food Funct. 2017 Nov 15;8(11):4139-4149. doi: 10.1039/c7fo01183k. PMID 29099521